CLINICAL TRIAL: NCT06042738
Title: The Impact of Antioxidant Food Supplementation on Seminal Antioxidant Capacity, Sperm DNA Fragmentation and Sperm Chromatin Quality in Subfertile Men With Oligoastenoteratozoospermia Randomized Clinical Trial
Brief Title: Investigation of The Effectiveness of Antioxidant Therapy in Oligoasthenoteratozoospermic Infertile Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Mesut Şengül, Principal investigator, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: OAT2023
Record Dates: First submitted 2023-07-25; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Male Infertility
Keywords: exercise; antioxidant; antioxidant capacity; sperm DNA fragmentation; protamine
MeSH Terms: conditions — Infertility, Male; Motor Activity

STUDY DESIGN:
Intervention Model Description: two groups with full (simple) randomization
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): group receiving antioxidant support
  Interventions: Combination Product: proxeed plus
- Group 2 (No Intervention): group that did not receive antioxidant support

INTERVENTIONS:
Combination Product: proxeed plus — Group 1 was recommended to receive a food supplement containing 2000 mg L-carnitine, 2000 mg fructose, 932 mg acetyl L-carnitine, 225 mg vitamin C, 115 mg citric acid, 50 mg coenzyme Q10, 14 mg zinc, 115 µg selenium, 3750 µg vitamin B12 and 500 µg folic acid as one sachet in the morning and evening
  Arms: Group 1

SUMMARY:
Approximately 30% of the factors that cause male infertility are due to idiopathic causes. Increased reactive oxygen species (ROS) due to many known and unknown factors cause male infertility by affecting spermatogenesis and sperm maturation. In this study, the effects of physical activity and antioxidant food supplementation on seminal antioxidant capacity, sperm DNA fragmentation index, sperm chromatin quality and sperm parameters were investigated in infertile cases.

DETAILED DESCRIPTION:
Material and Method: The study included subfertile men with idiopathic oligoasthenoteratozospermia seen at Ondokuz Mayıs University Faculty of Medicine between March 2021 and November 2021.

All subjects were recommended to do moderate physical activity for at least 45 minutes (at least 150 minutes-600 METs per week) 3-4 days a week for three months. A total of 48 cases were divided into two groups by computer-assisted (www.randomizer.org) complete (simple) randomization. In the first group (Group 1), 2000 mg L-carnitine, 2000 mg fructose, 932 mg acetyl L-carnitine, 225 mg vitamin C, 115 mg citric acid, 50 mg coenzyme Q10, 14 mg zinc, 115 µg selenium, 3750 µg Food supplement containing vitamin B12 and 500 µg folic acid was recommended as one sachet in the morning and evening, while antioxidant food supplement was not given to the second group (group 2). Before and after treatment, semen parameters, Hormone analyzes with ELISA method, physical activity evaluation with IPAQ questionnaire, seminal antioxidant capacity with Trolox equivalent antioxidant capacity (TEAC) measurement method, DNA fragmentation index with TUNEL method. and sperm chromatin structure was evaluated by aniline blue staining.

Student's t test was used for the variables showing normal distribution in independent groups, and Mann Whitney U test was used for the variables that did not fit the normal distribution. Paired t test was used for the variables showing normal distribution in the dependent groups, and Wilcoxon test was used for the variables that were found not to fit the normal distribution.

ELIGIBILITY:
Inclusion Criteria:

1) Clinical diagnosis of idiopathic oligoasthenoteratozoospermia

-

Exclusion Criteria:

1. Vasectomy
2. Azoospermia or severe oligozoospermia
3. Current use of a treatment or drug
4. Cancer, heart disease or cirrhosis history
5. Uncontrolled diabetes mellitus -

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Total Antioxidant Capacity | 3 months
  Total Antioxidant Capacity (TAC) was measured by the colorimetric assay using the antioxidant Assay Kit (Cayman Chemical, Michigan, USA). All seminal plasma samples were diluted prior to analysis. Standards were diluted sequentially. All samples and standards were placed in duplicate. Chromogen and metmyoglobin were added to both samples and standards. Hydrogen peroxide was added and then the plate was incubated. The absorbances of the standards and samples were measured at 750 nm using a microplate spectrophotometer (Multiscan GO, Thermo Scientific, Finland) after incubation.
  Calculations of each standard and sample were made to evaluate the assay. A standard Trolox curve was plotted with the mean absorbance of the standards. The TACs of the samples were calculated according to the formula using the linear regression of that standard curve and the average of the absorbance of samples: Antioxidant (mM) = [(Sample average absorbance) - (y-intercept)/ Slope] x Dilution
Sperm DNA Fragmentation | 3 months
  Sperm DNA Fragmentation (SDF) was analysed with TUNEL using the commercial In situ Cell Death Detection Kit. All samples were fixed with 4% paraformaldehyde (PFA). Fixed sperm samples were added onto polylysine-coated slides. Slides were kept in freshly prepared permeabilization solution on ice. For TUNEL reaction, label solution was mixed with enzyme solution, and 50 µl of the mix was dropped. Slides were incubated, afterward, they were washed three times and a mounting medium with DAPI was added. Samples were immediately examined and photographed using a fluorescent microscope. Photographs were analysed with the Image J program and at least 500 cells were evaluated from each sample. SDF was calculated as the number of sperm nuclei stained green as a percentage of the total sperm nuclei identified as blue in the same area.
% of histone-rich spermatozoa | 3 months
  Sperm pellets were washed then spread on clean slides and the smears were air dried. Dried smears were fixed with 3% glutaraldehyde and they were immersed in a 5% aniline blue solution in 4% glacial acetic acid. After staining, 200 sperm were counted at least on each slide at 1000x magnification at a light microscope. Pale blue spermatozoa that received less or no staining were considered protamine-rich, and spermatozoa partially or completely stained dark blue were evaluated as histone-rich.

CONTACTS AND LOCATIONS:
Overall Officials: Ramazan Asci, Study Director — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayıs University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sengul M, Hekim N, Asci R, Gunes S. The impact of antioxidants on antioxidant capacity, DNA fragmentation, and chromatin quality in subfertile men: a randomized clinical trial study. Rev Assoc Med Bras (1992). 2024 Nov 11;70(10):e20240211. doi: 10.1590/1806-9282.20240211. eCollection 2024. PMID 39536246

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Study Protocol and Statistical Analysis Plan (2021-03-16): https://cdn.clinicaltrials.gov/large-docs/38/NCT06042738/Prot_SAP_000.pdf
  • Study Protocol: Approval of Ethical Comittee (2021-03-16): https://cdn.clinicaltrials.gov/large-docs/38/NCT06042738/Prot_001.pdf